CLINICAL TRIAL: NCT04835974
Title: Metabolic Profile as a Predictor of No-reflow in Diabetic Patients Treated With Primary Percutaneous Coronary Intervention (PCI)
Brief Title: the No-reflow in Diabetic Patients Treated With Primary Percutaneous Coronary Intervention (PCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El Zahraa Gamal, Metabolic profile as a predictor of no reflow in diabetic patients treated with primary Percutaneous Coronary Intervention (PCI) ., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: No-reflow phenomenon
Record Dates: First submitted 2021-03-23; First posted 2021-04-08 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: No-Reflow Phenomenon
MeSH Terms: conditions — No-Reflow Phenomenon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diabetic patients with reflow phenomenon (Experimental): All Assiut University heart Hospital patients ,and who meet the listed inclusion and exclusion criteria will be eligible for the study. Patients' charts will be retrieved based on their intervention procedures. The charts will be reviewed and eligible patients will be filtered. The needed variables will be entered into our data base for later data analysis.
  Interventions: Diagnostic Test: 1- LDL-C (low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotein cholesterol) Ratio. 2- Glycemia will be assessed : RBS ( random blood sugar ) . 3- S

INTERVENTIONS:
Diagnostic Test: 1- LDL-C (low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotein cholesterol) Ratio. 2- Glycemia will be assessed : RBS ( random blood sugar ) . 3- S — Blood samples were obtained before PCI, and the following parameters will be measured:
  1. LDL-C (low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotein cholesterol) Ratio.
  2. Glycemia will be assessed : RBS ( random blood sugar ) .
  3. Serum Uric acid : S .UA

SUMMARY:
1- to find metabolic factors that correlate with the development of no reflow phenomenon that may help prevent its occurrence .

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) with its accompanying adverse sequelae is one of the most common causes of morbidity and mortality in the world .

Although reperfusion techniques for ST- elevation myocardial infarction (STEMI ) are constantly improving, no-reflow can still lead to poor prognosis .

At present, the exact mechanism of no-reflow remains unclear, but clinical and laboratory findings suggest that it is related to the embolism of the capillary bed, ischemic injury, vascular endothelial dysfunction, production of oxygen free radical , and other factors .

The no-reflow phenomenon is one of complications of poor functional and clinical outcomes for patients with (AMI) .

The no-reflow phenomenon is present in 25% to 30% of patients with (AMI) underwent successful coronary recanalization, as shown by angiography . The myocardial no-reflow phenomenon is associated with a reducution of antegrade myocardial blood flow inspite of an open infarct-related artery in patients with (STEMI ) undergoing (PCI). Importantly, no-reflow is known to be related to unfavorable clinical outcome and prognosis . The cause of this complex phenomenon is the variable combination of four pathogenetic components: distal atherothrombotic embolization, ischemic injury, reperfusion injury and susceptibility of coronary microcirculation to injury . As a consequence, appropriate strategies are expected to prevent or treat these components are expected to avoid the no-reflow. Coronary reperfusion therapy is widely performed in patients with (AMI) . However, in spite of patency of the infarct-related artery , there is no guarantee of salvage of myocardium at risk of ischemia .The no-reflow phenomenon is found in >30% of patients after thrombolysis or catheter-based (PCI) for (AMI) . It is important, therefore, to be able to predict which lesions are high risk for no reflow before beginning PCI .

There are numerous recognized risk factors for the development of coronary artery disease (CAD), one of the best known is the association between blood lipids and CAD . Several prospective studies have established that the risk of cardiac morbidity and mortality is directly related to the concentration of plasma cholesterol. ' The most prevalent view is that the increased risk of myocardial infarction associated with elevated plasma cholesterol levels can be adequately explained on the basis of the increase in number and severity of coronary atherosclerotic vascular lesions . .

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with STEMI treated with primary PCI

Exclusion Criteria:

non diabetic . with selected PCI

* (1) a history of an unprotected left main artery with severe liver and kidney diseases or coronary artery bypass grafting .

  (2) patients who had valvular disease or cardiomyopathy . (3) severe dissection, thromboembolism in other parts, or vasospasm; and known malignancy .

  (4) patients with contraindications for anticoagulant therapy, such as active visceral hemorrhage, hemorrhagic stroke, or ischemic stroke within half a year (including transient ischemic attack), or aortic dissection, or patients with hematological diseases complicated with coagulation disorders .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
measure serum random blood sugar | baseline
  to detect the correlation between the diabetus mellitus (serum random blood sugar) and no-reflow phenomenon and analysis of this metabolic factors in patient withSTEMI who will undergo primaru PCI and show its effects on no-reflow phenomenon that may help prevent its occurrence .

SECONDARY OUTCOMES:
measure the serum uric acid | baseline
  to detect the correlation between the serum uric acid , lipid profile and no-reflow phenomenon and show other metabolic factors effects on no-reflow to avoid its occurance
measure the lipid profile | baseline
  to detect the correlation between lipid profile and no-reflow phenomenon

REFERENCES:
- [Background] Bernstein JM, Lee J, Conboy K, Ellis E, Li P. The role of IgE mediated hypersensitivity in recurrent otitis media with effusion. Am J Otol. 1983 Jul;5(1):66-9. No abstract available. PMID 6683937